CLINICAL TRIAL: NCT04897971
Title: Use of MENSA to Improve the Diagnosis of Causative Infectious Agent and Monitor Infection Recovery in Orthopedic Spine Infection
Brief Title: Serum Based Diagnosis of and Monitoring of Infection Recovery in Orthopedic Spine Implant Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2946
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Staphylococcus Aureus Infection; Surgical Site Infection; Orthopedic Procedures; Spine
Keywords: Spine, Orthopedic Implant infection
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. No more than two, 1-gram (~ 2 cm3, total) pieces of surgical discard tissue will be collected from the area around the orthopedic implants.
  2. 5-10 mL of whole blood drawn into a 10 mL heparinized collection tube fort he purpose of collecting peripheral blood mono nuclear cells.
  3. 1-2 mL of whole blood drawn for preparing serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spine implant associated infection cohort: Adult patients undergoing revision spine surgeries with suspected infection of previous instrumentation.
  Interventions: Diagnostic Test: Medium enriched for newly synthesized antibodies in spine infection

INTERVENTIONS:
Diagnostic Test: Medium enriched for newly synthesized antibodies in spine infection — Medium enriched for newly synthesized antibodies titers in patients with Staphylococcus aureus infections of orthopedic spine implants at baseline and in the post operative period

SUMMARY:
The goal of this study is to test a new way to diagnose and track treatment of spine infections caused by the bacteria Staphylococcus aureus.

DETAILED DESCRIPTION:
Ongoing Staphylococcus aureus (S. aureus) infections of the spine associated with orthopedic hardware implants elicit prominent immune responses against a repertoire of proteins characteristic of the invading pathogen. Antibodies specific for these antigens can be measured in the serum or in a novel sample created by culturing circulating Antibody Secreting Cells (ASC) in vitro where they create an analytic fluid called here "medium enriched for newly synthesized antibodies" (MENSA). The hypothesis of this study addresses three essential attributes of this analytic approach that can yield both a valuable tool for research on spinal infections and in the future, this can be developed a clinical tool for diagnosis and monitoring of therapeutic success in patients. By measuring the emergence of these signature antibodies in the serum and/or MENSA, the goals of this study are: 1) To differentiate between patients with an ongoing S. aureus infections, not just "general infection, in the spine using only blood samples; 2) To track the success (or failure) of therapeutic interventions; and 3) to distinguish spinal infections from S. aureus infections in other sites by the repertoire of antibodies that are elicited.

ELIGIBILITY:
Inclusion Criteria:

* patients with known or suspected spinal infections associated with spinal orthopedic implant(s);
* patients over 18 years of age and younger than 85;
* patients undergoing spinal revision surgery.

Exclusion Criteria:

* Diagnosed as immuno-compromised or immuno-suppressed based on medication use;
* On-going or previously diagnosed musculoskeletal infections associated non-spine hardware (e.g., prosthetic hip, prosthetic knee, prosthetic shoulder);
* Current diabetic foot ulcer/infection;
* Patients undergoing cancer treatment (including radiation and chemotherapies);
* Pregnancy;
* Absence of a spleen;
* Over the age of 85 or under the age of 18.
* Weigh less than 110 pounds, or for which it would otherwise be unsafe for them to undergo a blood draw.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision spine surgeries at the University of Colorado Hospital. with suspected infection of previous instrumentation will be offered enrollment. The enrolled patients will be identified prior to surgery by the surgeons and research staff through radiographs and images contained in the medical records and the parameters of suspected infection which include:
  * Blood biomarkers: elevated C-reactive protein (CRP) and ESR (erythrocyte sedimentation rate), and white blood cell count
  * X-ray imaging: to show osteolysis and possibly implant-loosening
  * MRI or CT imaging: looking for fluid accumulations, evidence of inflammation, enhancements.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of Staphylococcus aureus spine implant associated infections correctly identified by "medium enriched for newly synthesized antibodies" (MENSA) | Baseline
  "A medium enriched for newly synthesized antibodies" (MENSA) is the supernatant collected from cultured antibody secreting cells. Peripheral blood monocytes (PBMCs) are washed and placed into cell culture. After 24 hours, the media contains a high concentration of newly made antibodies. This media is referred to as MENSA. This is tested to see if the antibodies collected react against a panel of antigens. MENSA immunoglobulin G (IgG) titers for each antigen will be assessed for their predictive ability to identify the presence of S. aureus in spine implant-associated infections using receiver operating characteristic (ROC) curve analysis (alone or in combination), with overall prediction accuracy summarized by the area-under-the-curve (AUC). Participants will then be categorized as Staphylococcus aureus (S. aureus) positive or negative based on MENSA. The percentage of correctly identified S. aureus determinations compared to clinical diagnosis will be determined.
Change "Medium enriched for newly synthesized antibodies" (MENSA) titers in the post-operative period | 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years post-surgery
  MENSA IgG titers (as defined in Outcome 1) will be measured at 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years post-surgery. A longitudinal measure of antibody activity defined as the average change per study visit from baseline will used to track infection clearance versus persistent infection. Levels of anti-S. aureus antibodies in MENSA should decline to background in patients whose infections have been successfully treated and remain elevated in those whose infections persist.
"Medium enriched for newly synthesized antibodies" (MENSA) titers in spine implant infections compared to S. aureus infections of other orthopedic site infections. | Baseline
  MENSA IgG titers (as defined in Outcome 1) will be compared to responses measured in a pre-existing collection of samples from patients who had experienced: 1) prosthetic joint infections; 2) septic arthritis; 3) diabetic foot infections; 4) soft-tissue infections; and 5) fracture-related infections. The goal will be to identify a combination of antigens that is uniquely discriminatory for spine infections.

SECONDARY OUTCOMES:
Confirmation of Staphylococcus aureus in spine implant associated infection by polymerase chain reaction (PCR) | Baseline
  Total DNA will be collected from surgical discarded tissue from sites adjacent to the infection. polymerase chain reaction (PCR) using primers that amplify a region of the Staphylococcus aureus genome will be run to confirm the presence/absence of Staphylococcus aureus at the infection site.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Ackert-Bicknell, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Univeristy of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muthukrishnan G, Soin S, Beck CA, Grier A, Brodell JD Jr, Lee CC, Ackert-Bicknell CL, Lee FE, Schwarz EM, Daiss JL. A Bioinformatic Approach to Utilize a Patient's Antibody-Secreting Cells against Staphylococcus aureus to Detect Challenging Musculoskeletal Infections. Immunohorizons. 2020 Jun 22;4(6):339-351. doi: 10.4049/immunohorizons.2000024. PMID 32571786
- [Background] Oh I, Muthukrishnan G, Ninomiya MJ, Brodell JD Jr, Smith BL, Lee CC, Gill SR, Beck CA, Schwarz EM, Daiss JL. Tracking Anti-Staphylococcus aureus Antibodies Produced In Vivo and Ex Vivo during Foot Salvage Therapy for Diabetic Foot Infections Reveals Prognostic Insights and Evidence of Diversified Humoral Immunity. Infect Immun. 2018 Nov 20;86(12):e00629-18. doi: 10.1128/IAI.00629-18. Print 2018 Dec. PMID 30275008
- [Background] Nishitani K, Beck CA, Rosenberg AF, Kates SL, Schwarz EM, Daiss JL. A Diagnostic Serum Antibody Test for Patients With Staphylococcus aureus Osteomyelitis. Clin Orthop Relat Res. 2015 Sep;473(9):2735-49. doi: 10.1007/s11999-015-4354-2. Epub 2015 May 27. PMID 26013151